CLINICAL TRIAL: NCT02423434
Title: Multinational Collaborative Evaluation of Corneal Confocal Microscopy as a Surrogate Endpoint for the Identification and Prediction of Diabetic Neuropathy in Type 1 Diabetes
Brief Title: Evaluation of Corneal Confocal Microscopy for the Identification and Prediction of Neuropathy in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Calgary (Other); Queensland University of Technology (Other); University of Michigan (Other); University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: DP3DK104386 (NIH); 1DP3DK104386-01 (NIH)
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Diabetic Polyneuropathy; Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Complications
Keywords: Corneal Confocal Microscopy; Diabetes Mellitus; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus; Diabetic Neuropathy; Diabetes Complications
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Corneal Confocal Microscopy subjects
  Interventions: Other: Exposure: Corneal nerve fibre morphology by the CCM Procedure

INTERVENTIONS:
Other: Exposure: Corneal nerve fibre morphology by the CCM Procedure — CCM is a non-invasive method for direct visualization of corneal nerve fibers. Previous research work has confirmed that corneal nerves status correlates with both small and large fibre damage as assessed by quantitative sensory testing and nerve conduction.
  In the current trial subjects will undergo a bilateral examination of the Bowman's layer of the cornea using the Rostock Cornea Module of the Heidelberg Tomograph III (Heidelberg Engineering, Smithfield RI, USA) to determine their corneal nerve fiber length, corneal nerve fiber density, corneal nerve branch density, and the tortuosity coefficient. Topical anaesthetic and a viscous gel medium will be applied to the eye, which will create a visual gel bridge between the cornea and the sterile single-use cap on the microscope objective lens. After the interface between the corneal epithelium and Bowman's layer is identified, batches of images will be taken and the most technically sound images will be identified and analyzed.

SUMMARY:
Through the multinational pooled dataset approach, this trial will aim to derive and validate specific in vivo Corneal Confocal Microscopy (CCM) parameter thresholds for the identification of diabetic polyneuropathy, and - more importantly - the identification of individuals at future risk. Results of the study will permit application in clinical practice and intervention trials for diabetic polyneuropathy (DPN) risk stratification.

The primary goal of the study is to re-examine individuals with type 1 and type 2 diabetes with and without neuropathy, who had CCM performed in the past as a part of their neurological examination, to assess concurrent and predictive validity of different CCM parameters in individuals . These subjects will be invited to the study to be re-examined by CCM along with other neurological tests (physical exam, nerve conduction studies, quantitative sensory testing, blood test and in some centres also skin biopsy) during the single study visit. Additionally CCM data will be analyzed both manually and by recently developed automated analytical software to evaluate accuracy of the automated method. Evaluation of automated image analysis will influence likelihood of successful knowledge translation of this surrogate biomarker for DPN into clinical practice - in which the procedure could be harmonized with annual retinal examinations - and into intervention trials.

Secondary aim of the study is to determine the factors associated with CCM parameters and their longitudinal change and collect bio-samples for future research in this field.

DETAILED DESCRIPTION:
The diffuse injury to peripheral nerves (diabetic neuropathy) is exceptionally common in type 1 diabetes, but there is a lack of an objective surrogate marker to identify early subclinical stages when treatments might be most effective, prior to late-stage progression to troublesome and costly foot infection, ulceration, and limb amputation. In contrast to the ability to objectively measure disease-specific surrogate markers for retinopathy and nephropathy, this lack of a diabetic neuropathy surrogate marker has seriously impeded the development of specific interventions in clinical research trials. Representing 5 independent research groups that have together created a consortium of investigators dedicated to the development of a surrogate marker for early diabetic neuropathy, we have focused on using the eye as a window to non-invasively image by a method of in-vivo corneal confocal microscopy (CCM) the small nerve fibres that innervate the cornea. We have demonstrated that changes in these nerve fibre endings occur early in the development of neuropathy, reflect well the changes seen in other peripheral nerves by invasive skin biopsy evaluation, and that their measurement is feasible and reproducible. As a multinational consortium, we have the benefit in this proposal of pooling multiple cohorts to apply the most valid study methods in biomarker development. First, we aim to determine in the analysis of an existing pooled dataset of 516 type 1 and 524 type 2 diabetes subjects the exact levels of CCM measurement that can identify the presence of diabetic neuropathy. Secondly, we propose over three years to re-examine at least 70% of this cohort, which will provide 5- to 7-year follow-up data to determine which type and level of CCM measurement can predict the future onset of neuropathy, as well as its progression in those who had neuropathy at baseline. Finally, we will evaluate the role of time- and cost-saving automated image analysis software. By virtue of large sample size from data pooling, we are uniquely afforded the methodological power to confirm our objectives by way of separate derivation and validation analysis sets. Through a unique and unprecedented multinational pooled dataset approach for diabetic neuropathy, this work will derive and validate specific CCM parameter thresholds for the identification of neuropathy, and - more importantly - the identification of individuals at future risk. These results will permit application in clinical practice and intervention trials for neuropathy risk stratification. Evaluation of automated image analysis will influence likelihood of successful knowledge translation of this surrogate biomarker into clinical practice - in which the procedure could be harmonized with annual retinal examinations - and into intervention trials.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of any gender or race aged 18 or above
* Type 1 diabetes mellitus or type 2 diabetes mellitus as defined by the American Diabetes Association guidelines (2014) of any duration
* Availability of the initial CCM examination performed two to eight years ago
* Ability to understand and cooperate with study procedures

Exclusion Criteria:

* Confirmed to have neuropathy owing to non-diabetic causes (such as familial, alcoholic, nutritional, uremic)
* Current eye infection, corneal damage, or severe movement disorders which could preclude a safe CCM exam
* Allergy to proparacaine (the ocular topical anaesthetic used for the CCM exam)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This longitudinal observational cohort study of diagnosis involves follow-up in two study groups:
  A. Five- to seven-year follow-up re-examination of 5 well-characterized type 1 diabetes (T1D) cohorts (N=516) comprising a neuropathic subset and a non-neuropathic subset.
  B. Three- to six-year follow-up re-examination of 4 well-characterized type 2 diabetes (T2D) cohorts (N=524) each comprising a neuropathic subset and a non-neuropathic subset.
  T1D Subjects. The five study sites are composed of cohort studies for T1D initiated between 2008 and 2011. Together, the five sites have studied 516 subjects at baseline with T1D, 363 without DPN and 151 with DPN at baseline.
  T2D Subjects. Four of the sites have studied subjects with T2D. Together, the four sites have studied 524 subjects at baseline with T2D, 241 without DPN and 283 with DPN at baseline.
  Of the 1040 total subjects examined in baseline procedures, we anticipate follow-up of 70% for a total re-examined cohort 729.
Sampling Method: Non-Probability Sample
Enrollment: 624 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the Concurrent Validity of CCM Parameters from Cross-Sectional Analysis of Well-Characterized T1D and T2D Subjects. | Any data obtained from pre-study measurements
Evaluate the Predictive Validity of CCM Parameters based on the 5-7 year Incidence of Neuropathy in Well-Characterized T1D and T2D Subjects Without Neuropathy at Baseline | Study visit
Evaluate the Predictive Validity of CCM Parameters for 5-7 year Progression of Neuropathy | Study visit
Comparison of Manual versus Automated Image analysis | Pre-study and study visit data

SECONDARY OUTCOMES:
Determination of the Factors associated with CCM Parameters and their Longitudinal Change | Study visit

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Perkins, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (5):
- University of Michigan, Ann Arbor, Michigan, United States
- Queensland University of Technology, Brisbane, Australia
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Mount Sinai Hospital and University Health Network, Toronto, Ontario
- University of Manchester, Manchester, United Kingdom

REFERENCES:
- [Background] Tavakoli M, Ferdousi M, Petropoulos IN, Morris J, Pritchard N, Zhivov A, Ziegler D, Pacaud D, Romanchuk K, Perkins BA, Lovblom LE, Bril V, Singleton JR, Smith G, Boulton AJ, Efron N, Malik RA. Normative values for corneal nerve morphology assessed using corneal confocal microscopy: a multinational normative data set. Diabetes Care. 2015 May;38(5):838-43. doi: 10.2337/dc14-2311. Epub 2015 Jan 29. PMID 25633665
- [Background] Pritchard N, Edwards K, Russell AW, Perkins BA, Malik RA, Efron N. Corneal confocal microscopy predicts 4-year incident peripheral neuropathy in type 1 diabetes. Diabetes Care. 2015 Apr;38(4):671-5. doi: 10.2337/dc14-2114. Epub 2015 Jan 8. PMID 25573881
- [Background] Tavakoli M, Begum P, McLaughlin J, Malik RA. Corneal confocal microscopy for the diagnosis of diabetic autonomic neuropathy. Muscle Nerve. 2015 Sep;52(3):363-70. doi: 10.1002/mus.24553. Epub 2015 Jun 18. PMID 25556884
- [Background] Dehghani C, Pritchard N, Edwards K, Vagenas D, Russell AW, Malik RA, Efron N. Natural history of corneal nerve morphology in mild neuropathy associated with type 1 diabetes: development of a potential measure of diabetic peripheral neuropathy. Invest Ophthalmol Vis Sci. 2014 Nov 18;55(12):7982-90. doi: 10.1167/iovs.14-15605. PMID 25406279
- [Background] Maddaloni E, Sabatino F, Del Toro R, Crugliano S, Grande S, Lauria Pantano A, Maurizi AR, Palermo A, Bonini S, Pozzilli P, Manfrini S. In vivo corneal confocal microscopy as a novel non-invasive tool to investigate cardiac autonomic neuropathy in Type 1 diabetes. Diabet Med. 2015 Feb;32(2):262-6. doi: 10.1111/dme.12583. Epub 2014 Sep 24. PMID 25251450
- [Background] Stem MS, Hussain M, Lentz SI, Raval N, Gardner TW, Pop-Busui R, Shtein RM. Differential reduction in corneal nerve fiber length in patients with type 1 or type 2 diabetes mellitus. J Diabetes Complications. 2014 Sep-Oct;28(5):658-61. doi: 10.1016/j.jdiacomp.2014.06.007. Epub 2014 Jun 17. PMID 25044236
- [Background] Asghar O, Petropoulos IN, Alam U, Jones W, Jeziorska M, Marshall A, Ponirakis G, Fadavi H, Boulton AJ, Tavakoli M, Malik RA. Corneal confocal microscopy detects neuropathy in subjects with impaired glucose tolerance. Diabetes Care. 2014 Sep;37(9):2643-6. doi: 10.2337/dc14-0279. Epub 2014 Jun 26. PMID 24969581
- [Background] Edwards K, Pritchard N, Vagenas D, Russell A, Malik RA, Efron N. Standardizing corneal nerve fibre length for nerve tortuosity increases its association with measures of diabetic neuropathy. Diabet Med. 2014 Oct;31(10):1205-9. doi: 10.1111/dme.12466. Epub 2014 May 24. PMID 24750318
- [Background] Ziegler D, Papanas N, Zhivov A, Allgeier S, Winter K, Ziegler I, Bruggemann J, Strom A, Peschel S, Kohler B, Stachs O, Guthoff RF, Roden M; German Diabetes Study (GDS) Group. Early detection of nerve fiber loss by corneal confocal microscopy and skin biopsy in recently diagnosed type 2 diabetes. Diabetes. 2014 Jul;63(7):2454-63. doi: 10.2337/db13-1819. Epub 2014 Feb 26. PMID 24574045
- [Background] Petropoulos IN, Alam U, Fadavi H, Marshall A, Asghar O, Dabbah MA, Chen X, Graham J, Ponirakis G, Boulton AJ, Tavakoli M, Malik RA. Rapid automated diagnosis of diabetic peripheral neuropathy with in vivo corneal confocal microscopy. Invest Ophthalmol Vis Sci. 2014 Apr 3;55(4):2071-8. doi: 10.1167/iovs.13-13787. PMID 24569580
- [Background] Tavakoli M, Petropoulos IN, Malik RA. Corneal confocal microscopy to assess diabetic neuropathy: an eye on the foot. J Diabetes Sci Technol. 2013 Sep 1;7(5):1179-89. doi: 10.1177/193229681300700509. PMID 24124944
- [Background] Petropoulos IN, Alam U, Fadavi H, Asghar O, Green P, Ponirakis G, Marshall A, Boulton AJ, Tavakoli M, Malik RA. Corneal nerve loss detected with corneal confocal microscopy is symmetrical and related to the severity of diabetic polyneuropathy. Diabetes Care. 2013 Nov;36(11):3646-51. doi: 10.2337/dc13-0193. Epub 2013 Jul 22. PMID 23877983
- [Background] Papanas N, Ziegler D. Corneal confocal microscopy: a new technique for early detection of diabetic neuropathy. Curr Diab Rep. 2013 Aug;13(4):488-99. doi: 10.1007/s11892-013-0390-z. PMID 23666893
- [Background] Sivaskandarajah GA, Halpern EM, Lovblom LE, Weisman A, Orlov S, Bril V, Perkins BA. Structure-function relationship between corneal nerves and conventional small-fiber tests in type 1 diabetes. Diabetes Care. 2013 Sep;36(9):2748-55. doi: 10.2337/dc12-2075. Epub 2013 Apr 11. PMID 23579181
- [Background] Halpern EM, Lovblom LE, Orlov S, Ahmed A, Bril V, Perkins BA. The impact of common variation in the definition of diabetic sensorimotor polyneuropathy on the validity of corneal in vivo confocal microscopy in patients with type 1 diabetes: a brief report. J Diabetes Complications. 2013 May-Jun;27(3):240-2. doi: 10.1016/j.jdiacomp.2012.10.011. Epub 2012 Dec 21. PMID 23266297
- [Background] Shtein RM, Callaghan BC. Corneal confocal microscopy as a measure of diabetic neuropathy. Diabetes. 2013 Jan;62(1):25-6. doi: 10.2337/db12-1114. No abstract available. PMID 23258907
- [Background] Efron N. Assessing diabetic neuropathy using corneal confocal microscopy. Invest Ophthalmol Vis Sci. 2012 Dec 7;53(13):8075. doi: 10.1167/iovs.12-11308. No abstract available. PMID 23221463
- [Background] Tavakoli M, Petropoulos IN, Malik RA. Assessing corneal nerve structure and function in diabetic neuropathy. Clin Exp Optom. 2012 May;95(3):338-47. doi: 10.1111/j.1444-0938.2012.00743.x. PMID 22594548
- [Background] Wu T, Ahmed A, Bril V, Orszag A, Ng E, Nwe P, Perkins BA. Variables associated with corneal confocal microscopy parameters in healthy volunteers: implications for diabetic neuropathy screening. Diabet Med. 2012 Sep;29(9):e297-303. doi: 10.1111/j.1464-5491.2012.03678.x. PMID 22519850
- [Background] Ahmed A, Bril V, Orszag A, Paulson J, Yeung E, Ngo M, Orlov S, Perkins BA. Detection of diabetic sensorimotor polyneuropathy by corneal confocal microscopy in type 1 diabetes: a concurrent validity study. Diabetes Care. 2012 Apr;35(4):821-8. doi: 10.2337/dc11-1396. Epub 2012 Feb 8. PMID 22323412
- [Background] Dabbah MA, Graham J, Petropoulos IN, Tavakoli M, Malik RA. Automatic analysis of diabetic peripheral neuropathy using multi-scale quantitative morphology of nerve fibres in corneal confocal microscopy imaging. Med Image Anal. 2011 Oct;15(5):738-47. doi: 10.1016/j.media.2011.05.016. Epub 2011 Jun 13. PMID 21719344
- [Background] Tavakoli M, Kallinikos P, Iqbal A, Herbert A, Fadavi H, Efron N, Boulton AJ, A Malik R. Corneal confocal microscopy detects improvement in corneal nerve morphology with an improvement in risk factors for diabetic neuropathy. Diabet Med. 2011 Oct;28(10):1261-7. doi: 10.1111/j.1464-5491.2011.03372.x. PMID 21699561
- [Background] Malik RA, Veves A, Tesfaye S, Smith G, Cameron N, Zochodne D, Lauria G; Toronto Consensus Panel on Diabetic Neuropathy. Small fibre neuropathy: role in the diagnosis of diabetic sensorimotor polyneuropathy. Diabetes Metab Res Rev. 2011 Oct;27(7):678-84. doi: 10.1002/dmrr.1222. PMID 21695760
- [Background] Hertz P, Bril V, Orszag A, Ahmed A, Ng E, Nwe P, Ngo M, Perkins BA. Reproducibility of in vivo corneal confocal microscopy as a novel screening test for early diabetic sensorimotor polyneuropathy. Diabet Med. 2011 Oct;28(10):1253-60. doi: 10.1111/j.1464-5491.2011.03299.x. PMID 21434993
- [Background] Pritchard N, Edwards K, Shahidi AM, Sampson GP, Russell AW, Malik RA, Efron N. Corneal markers of diabetic neuropathy. Ocul Surf. 2011 Jan;9(1):17-28. doi: 10.1016/s1542-0124(11)70006-4. PMID 21338566
- [Background] Efron N, Edwards K, Roper N, Pritchard N, Sampson GP, Shahidi AM, Vagenas D, Russell A, Graham J, Dabbah MA, Malik RA. Repeatability of measuring corneal subbasal nerve fiber length in individuals with type 2 diabetes. Eye Contact Lens. 2010 Sep;36(5):245-8. doi: 10.1097/ICL.0b013e3181eea915. PMID 20724854
- [Background] Messmer EM, Schmid-Tannwald C, Zapp D, Kampik A. In vivo confocal microscopy of corneal small fiber damage in diabetes mellitus. Graefes Arch Clin Exp Ophthalmol. 2010 Sep;248(9):1307-12. doi: 10.1007/s00417-010-1396-8. Epub 2010 May 21. PMID 20490534
- [Background] Tavakoli M, Quattrini C, Abbott C, Kallinikos P, Marshall A, Finnigan J, Morgan P, Efron N, Boulton AJ, Malik RA. Corneal confocal microscopy: a novel noninvasive test to diagnose and stratify the severity of human diabetic neuropathy. Diabetes Care. 2010 Aug;33(8):1792-7. doi: 10.2337/dc10-0253. Epub 2010 Apr 30. PMID 20435796
- [Background] Midena E, Brugin E, Ghirlando A, Sommavilla M, Avogaro A. Corneal diabetic neuropathy: a confocal microscopy study. J Refract Surg. 2006 Nov;22(9 Suppl):S1047-52. doi: 10.3928/1081-597X-20061102-08. PMID 17444092
- [Background] Mocan MC, Durukan I, Irkec M, Orhan M. Morphologic alterations of both the stromal and subbasal nerves in the corneas of patients with diabetes. Cornea. 2006 Aug;25(7):769-73. doi: 10.1097/01.ico.0000224640.58848.54. PMID 17068451
- [Background] Hossain P, Sachdev A, Malik RA. Early detection of diabetic peripheral neuropathy with corneal confocal microscopy. Lancet. 2005 Oct 15-21;366(9494):1340-3. doi: 10.1016/S0140-6736(05)67546-0. No abstract available. PMID 16226599
- [Background] Kallinikos P, Berhanu M, O'Donnell C, Boulton AJ, Efron N, Malik RA. Corneal nerve tortuosity in diabetic patients with neuropathy. Invest Ophthalmol Vis Sci. 2004 Feb;45(2):418-22. doi: 10.1167/iovs.03-0637. PMID 14744880
- [Background] Malik RA, Kallinikos P, Abbott CA, van Schie CH, Morgan P, Efron N, Boulton AJ. Corneal confocal microscopy: a non-invasive surrogate of nerve fibre damage and repair in diabetic patients. Diabetologia. 2003 May;46(5):683-8. doi: 10.1007/s00125-003-1086-8. Epub 2003 May 9. PMID 12739016